CLINICAL TRIAL: NCT05102032
Title: Impact of a Minimally Invasive Approach to Laparoscopic Hysterectomy on Postoperative Recovery
Acronym: MIN-HYSTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANEST-01-2019
Record Dates: First submitted 2019-10-03; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Uterus Disease
Keywords: post operative recovery; laparoscopic hysterectomy; mini invasive surgery; low pressure laparoscopy
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional approach (Active Comparator): Conventional approach to laparoscopic hysterectomy
  Interventions: Procedure: Conventional approach
- Mini-invasive approach (Experimental): Mini-invasive approach to laparoscopic hysterectomy
  Interventions: Procedure: mini invasive approach

INTERVENTIONS:
Procedure: mini invasive approach — using mini-trocars (3 trocars of 3 mm and a 5 mm-optic trocar) with insufflation pressures of less than 8 mmHg.
  Arms: Mini-invasive approach
Procedure: Conventional approach — laparoscopic procedure including standard trocars (3 trocars of 5 mm and a 10 mm-optic trocar) with insufflation pressures between 10 and 12 mmHg.
  Arms: Conventional approach

SUMMARY:
Background Managing perioperative stress, including endocrino-metabolic changes and, inflammatory and pain responses, is a major challenge to improve patient's recovery. Currently, minimally invasive surgical procedures combined with multimodal analgesia are commonly used to increase the quality of postoperative period.

Purpose To demonstrate that a minimally invasive approach including low insufflation pressure and minitrocars in laparoscopic hysterectomy improves postoperative recovery and reduces pain stimulation and opioid consumption in comparison with a conventional approach.

Methods After informed consent, all patients scheduled for a laparoscopic hysterectomy including those with carcinologic disease will be part of this monocentric prospective randomized double-blinded study.

At admission in our outpatient unit, patients will have to fill the Post-operative Quality of Recovery Scale assessment form, before to be randomized into one of the following two groups:

* Conventional approach: laparoscopic procedure including standard trocars (3 trocars of 5 mm and a 10 mm-optic trocar) with insufflation pressures between 10 and 12 mmHg.
* Mini-invasive approach : laparoscopic surgery using mini-trocars (3 trocars of 3 mm and a 5 mm-optic trocar) with insufflation pressures of less than 8 mmHg.

Both groups will have general anesthesia with a deep neuromuscular blockade (TOF = 0 at the thumb adductor) and will benefit of our enhanced recovery program. Patients and evaluators will be blind regarding the allocated group.

The primary outcome is a comparison of the postoperative recovery between the two groups through the Post-operative Quality of Recovery Scale.This evaluation will include pain data, nausea/vomiting evaluation and cognitive function 6 hours after surgery.

Secondary outcomes are morphine consumption surgical comfort and patient satisfaction.

DETAILED DESCRIPTION:
Introduction About 43,000 hysterectomies were performed in France in 2016 half of them as a laparoscopic procedure. Compared to vaginal hysterectomy, laparoscopic surgery decreases postoperative pain and hospital length of stay [PubMed ID: 25524534 ]. Laparoscopic hysterectomy is also the most common surgical technique in the USA within enhanced recovery after surgery programs (ERAS)[2]. However, postoperative pain is still an important issue and results in most of the early re-admissions [3]. In addition, control of intraoperative stress, including painful stimuli, but also endocrine-metabolic and inflammatory responses is a major component of patient's recovery improvement. Reducing length of stay can lead to a possible outpatient surgery with a high level of quality and safety.

Hysterectomy in outpatient setting is barely done in France (0.1% in 2012 and 1.5% in 2017) compare to USA (more than 50%) so there is still a significant scope of improvement [2].

Many parameters need to be controlled to reduce perioperative stress [4,5]. Francophone teams showed that the use of mini-invasive techniques such as low and stable abdominal insufflation pressure is an important factor regarding pain and inflammation after gynecological surgery [6,7]. Furthermore to reduce parietal and peritoneal injuries can be achieved by using very small trocars while allowing surgery to be performed in good conditions [8,9]. Some teams have combined these two techniques with promising results in abdominal surgery [10].

The choice of anesthesia technic within an ERAS program that include quick elimination drugs, vascular filling monitoring and optimization, prevention of hypothermia and postoperative nausea/vomiting (PONV), as well as a multimodal analgesia, including loco-regional analgesia allow a faster postoperative recovery after pelvic surgery [11, 12]. Among these parameters, post-operative pain management is a major component. It has been demonstrated that pain prolongs surgical stress, delays mobilization and full recovery. Opioid medication therapy results in many adverse effects (PONV, sedation) and delays postoperative recovery[12]. Furthermore, availability of opioids at home is currently a real public health issue[13]. After a conventional hysterectomy use of opioids is almost systematic[14]. Therefore the challenge is to provide effective analgesia with the minimum of opioids use. Anesthesia with a deep neuromuscular blockade allows a low peritoneal pressure while maintaining optimal surgical comfort[15].

Hypothesis A mini-invasive approach of laparoscopic hysterectomy, combining mini-trocars and low pneumoperitoneum pressure would improve quality of post-operative recovery and reduce length of stay in the hospital allowing the procedure to be performed as outpatient surgery.

Purposes

* Primary goal: to demonstrate that a mini-invasive laparoscopic hysterectomy compared to a conventional approach improves the PQRS score.
* Secondary goal:

To assess intraoperative pain intensity using the Analgesia Nociception Index (ANI) and whether minimally invasive surgery reduces the use of per- and postoperative opioids, PONV and patient satisfaction.

Methods This randomized prospective study will be carried out according to CONSORT methodological standards[17].

Information and recruitment During the pre-operative clinic, surgeon will check patient's eligibility regarding the inclusion criteria and patients will receive oral and written inform consent about the study. During anesthesia clinic, eligibility for ambulatory surgery will be confirmed and informed consent will be obtained. Throughout the duration of the study (24 hours), the patient will not be able to be included in any other research protocol that could affect her post-operative recovery.

Population After informed consent, all eligible patients undergoing laparoscopic hysterectomy surgery for benign or malignant affections will be included. Inclusion criteria are: stable ASA (American Society of Anesthesiologists )score <3, no contraindication to take nonsteroidal anti-inflammatory drugs , absence of chronic pain, perfect understanding of post-operative psycho-motor assessment, presence of an attendant, distance between home and hospital allowing a possible quick readmission and acceptance to respect all the given medical instructions.

Patients will be systematically excluded in case of laparo-conversion and surgical or anesthetic complication.

Randomization and PQRS assessment:

After admission in the day surgery unit all patient included in the study will fill a PQRS form before to be randomized in one of the two groups. Randomization and intraoperative patient care will not be achieved by the PQRS assessor.

Randomization into one of the two arms will be done by using a remote computer randomization system :

* Conv group conventional approach : laparoscopic surgery using standard trocars (3 trocars of 5 mm and a 10 mm-optic trocar) with insufflation pressures between 10 and 12 mmHg.
* Mini-inv group mini-invasive approach: laparoscopic surgery using mini-trocars (3 trocars of 3 mm and a 5 mm-optic trocar) with insufflation pressures of less than 8 mmHg.

Both group will have an anesthesia with a deep neuromuscular blockade (TOF = 0 at the thumb adductor).

Neither the patient nor the evaluator will be aware of the randomization group.

- The pre-operative and H6 PQRS score will be collected by an anesthesiologist not involve in patient care either per or post operatively up to 24h after surgery.

Perioperative management All patient will benefit of our ERAS protocol: fasting allowing the use of drinks up to 2 hours before anesthesia[16], general anesthesia with oro-tracheal intubation and protective mechanical ventilation (current tidal volume between 6-8 ml/kg of ideal weight and peep at 5 cmH2O) with a mixture of air and oxygen (50/50) and multimodal analgesia with intravenous lidocaine infusion (1,5 mg/kg bolus immediately after induction followed by a continuous infusion of 1,5 mg/kg/h stopped 20 min before the end of the procedure. Anesthesia will be performed according to our department protocol : induction and maintenance of anesthesia by propofol/remifentanil operated by target controlled intravenous anesthesia system (TIVA); anesthetic depth monitored with a bispectral index (BIS) between 45 and 55; per-operative analgesia provided by remifentanil with a brain concentration objective 0,35 ng/L for induction. Quality of analgesia will be monitored through the Analgesia Nociception Index (ANI). Remifentanil brain concentration objective will be changed to keep ANI in a range of 50 to 70. Depth of neuromuscular block with atracurium will be monitored by train-of-four. Neuromuscular blockade will be antagonized at the end of surgery according to the recommended procedure [17].

Routine analgesia will be started 20 minutes before the end of the procedure : paracetamol 1 g and ketoprofen up to 100 mg according to age and kidney function. Intraperitoneal (20 ml) and trocars orifices (10 ml) infiltration will be achieved by 2 mg/ml ropivacaine at the end of the procedure. In addition, heated blanket will be used to prevent hypothermia and central temperature will be monitored with esophageal temperature sensor. Dexamethasone 8 mg and droperidol 0.625 mg will be given to prevent PONV. Fluid therapy will be limited to 2 ml/kg/h besides blood loss compensation with a balanced solution of Ringer-Lactate. No urinary catheter will be placed.

In the Post-anesthesia care unit (PACU), pain at rest and cough will be assessed using a verbal numeric scale (VNS) between 0 (no pain) and 10 (worst pain imaginable). Patients will receive morphine intravenously (3 mg every 5 min) if the VNS level is >3/10. In the case of PONV, intravenous ondansetron 4 mg will be given.

Patients will be allowed to feed and intravenous catheter will be removed as soon as they leave the PACU. Patients will be invited to walk as soon as they can. Preventive anticoagulation with enoxaparin will be started 6 hours postoperatively. Postoperative analgesia will be managed by a combination of paracetamol 500 mg and opium 20 mg and ketoprofen 50 mg every 6 hours.

Patient will be discharged from the day surgery unit according to a "Chung score" > 9. Decision to keep the patient overnight will be made by the surgeon and anesthesiologist in charge of the patient regardless of the study or randomization group.

Twenty four hours after surgery, outpatient will be called at home and inpatient seen in her room by a research assistant to answer to a satisfaction survey and to assess postoperative pain intensity and by mouth morphine consumption.

Outcomes evaluation The primary outcome is a comparison between the two groups of immediate postoperative recovery as determined by the PQRS score [18], applied at the 6th postoperative hour (pain score, PONV and cognitive recovery).

The secondary outcomes are :

* intraoperative intensity of nociceptive stimulation measured by the intraoperative opioids consumption (remifentanil) according to the Analgesia Nociception Index (ANI) [19]
* postoperative pain intensity at rest, cough and walk (if possible) and based on the Verbal Numeric Scale (VNS) at H2, H6 and H24 post-operative, intravenous morphine consumption in PACU and by mouth opioids (morphine sulfate) during the first 24 post-operative hours
* Incidence of PONV
* Percentage of patients who reached the preoperative PQRS score at H6
* Surgical comfort on the Leiden scale [20]
* Surgery duration, length of stay in PACU (Aldrete score/15min)
* Number of patients with PADSS scores < 9 at H2 and H6 [21]
* Number of outpatients
* Bowel movement at H24 post-operative
* Number of patients who returned to hospital after discharge (or requiring medical contact) within 7 days after surgery.
* Patient satisfaction (EVAN score) [22]
* Potential adverse events

Statistical analysis The number of patients required to show a 5-point difference in the PQRS score, with a risk α of 5% and a risk β of 20%, taking into account a baseline score in the Conv group of 30 +/- 5 at H6 is 31 patients per group. With 20% of patients included but not evaluable or with deviations from protocol, 37 patients per group should be included. The statistical analysis will be carried out on a per-protocol basis and with intention to treat. It will be based on the t-Student test for the main criterion (PQRS) and Mann-Whitney or Chi-2 tests for other parameters depending on the type of parameter.

ELIGIBILITY:
Inclusion Criteria:

* programmed to laparoscopic hysterectomy
* stable ASA score <3
* no contraindication to take nonsteroidal anti-inflammatory drugs
* absence of chronic pain
* perfect understanding of post-operative psycho-motor assessment
* presence of an attendant
* distance between home and hospital allowing a possible quick readmission
* acceptance to respect all the given medical instructions.

Exclusion Criteria:

* laparo-conversion and surgical or anesthetic complication.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
immediate postoperative recovery | 6th post-operative hour
  determined by the Post Operative Quality of recovery scale PQRS (pain score, PONV and cognitive recovery)

SECONDARY OUTCOMES:
intraoperative intensity of nociceptive stimulation | 4th induction hour
  measured by the intraoperative opioids consumption (remifentanil) according to the Analgesia Nociception Index (ANI) in microgram.
postoperative pain intensity: Verbal Numeric Scale (VNS) | 2nd, 6th and 24th post-operatives hours
  measured at rest, cough and walk (if possible) and based on the Verbal Numeric Scale (VNS) from 0 to 10.
Patient satisfaction: EVAN G score | 24th post-operative hour
  EVAN G score.
rate of return after discharge | Day 7 after discharge
  % of patients who returned to hospital after discharge.
Bowel movement | Day 1 after discharge
  % of patients who had bowel movement in each group
Number of outpatients | Day 1 after discharge
  rate of outpatients (%)
PADSS scores | 2nd and 6th post-operatives hours
  rate of patients who had PADSS score <9.
Surgery duration, length of stay in PACU | 4th post-operative hour
  In hh:mn
Surgical comfort | 6th post-operative hour
  Leiden scale
intravenous morphine consumption | 2nd, 6th and 24th post-operatives hours
  measured in PACU and by mouth opioids in mg.
Incidence of PONV | 2nd, 6th and 24th post-operatives hours
  rate of patients with PONV

CONTACTS AND LOCATIONS:
Overall Officials: Karim BOUATTOUR, Doctor, Principal Investigator — Institut Mutualiste Montsouris
Locations (1):
- Insitut Mutualiste Montsouris, Paris, France

REFERENCES:
- [Background] Allam IS, Makled AK, Gomaa IA, El Bishry GM, Bayoumy HA, Ali DF. Total laparoscopic hysterectomy, vaginal hysterectomy and total abdominal hysterectomy using electrosurgical bipolar vessel sealing technique: a randomized controlled trial. Arch Gynecol Obstet. 2015 Jun;291(6):1341-5. doi: 10.1007/s00404-014-3571-3. Epub 2014 Dec 19. PMID 25524534
- [Background] Cohen SL, Ajao MO, Clark NV, Vitonis AF, Einarsson JI. Outpatient Hysterectomy Volume in the United States. Obstet Gynecol. 2017 Jul;130(1):130-137. doi: 10.1097/AOG.0000000000002103. PMID 28594764
- [Background] Penn CA, Morgan DM, Rice LW, Harris JA, Rauh-Hain JA, Uppal S. Timing of and Reasons for Unplanned 30-Day Readmission After Hysterectomy for Benign Disease. Obstet Gynecol. 2016 Oct;128(4):889-897. doi: 10.1097/AOG.0000000000001599. PMID 27607868
- [Background] Wijk L, Franzen K, Ljungqvist O, Nilsson K. Implementing a structured Enhanced Recovery After Surgery (ERAS) protocol reduces length of stay after abdominal hysterectomy. Acta Obstet Gynecol Scand. 2014 Aug;93(8):749-56. doi: 10.1111/aogs.12423. Epub 2014 Jun 13. PMID 24828471
- [Background] Wijk L, Franzen K, Ljungqvist O, Nilsson K. Enhanced Recovery after Surgery Protocol in Abdominal Hysterectomies for Malignant versus Benign Disease. Gynecol Obstet Invest. 2016;81(5):461-7. doi: 10.1159/000443396. Epub 2016 Jan 23. PMID 26799328
- [Background] Kyle EB, Maheux-Lacroix S, Boutin A, Laberge PY, Lemyre M. Low vs Standard Pressures in Gynecologic Laparoscopy: a Systematic Review. JSLS. 2016 Jan-Mar;20(1):e2015.00113. doi: 10.4293/JSLS.2015.00113. PMID 26955258
- [Background] Sroussi J, Elies A, Rigouzzo A, Louvet N, Mezzadri M, Fazel A, Benifla JL. Low pressure gynecological laparoscopy (7mmHg) with AirSeal(R) System versus a standard insufflation (15mmHg): A pilot study in 60 patients. J Gynecol Obstet Hum Reprod. 2017 Feb;46(2):155-158. doi: 10.1016/j.jogoh.2016.09.003. Epub 2017 Jan 30. PMID 28403972
- [Background] Carvalho GL, Paquentin EM, Redan JA, Shadduck PP. The Science Behind Mini-Laparoscopic Cholecystectomy. Surg Technol Int. 2016 Oct 26;29:93-98. PMID 27466870
- [Background] Redan JA, Humphries AR, Farmer B, Paquentin EM, Koh CH, Chung MK, Stringel G, McCarus SD, Carvalho G, Diaz RG, Shadduck PP. "Big Operations Using Mini Instruments": The Evolution of Mini Laparoscopy in the Surgical Realm. Surg Technol Int. 2015 Nov;27:19-30. PMID 26680376
- [Background] de'Angelis N, Petrucciani N, Giannandrea G, Brunetti F. The protocol of low-impact laparoscopic cholecystectomy: the combination of mini-laparoscopy and low-pressure pneumoperitoneum. Updates Surg. 2018 Dec;70(4):553-556. doi: 10.1007/s13304-018-0591-8. Epub 2018 Aug 29. PMID 30159821
- [Background] Lee WK, Kim MS, Kang SW, Kim S, Lee JR. Type of anaesthesia and patient quality of recovery: a randomized trial comparing propofol-remifentanil total i.v. anaesthesia with desflurane anaesthesia. Br J Anaesth. 2015 Apr;114(4):663-8. doi: 10.1093/bja/aeu405. Epub 2014 Dec 10. PMID 25500679
- [Background] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):801-16. doi: 10.1016/j.clnu.2012.08.012. Epub 2012 Sep 26. PMID 23062720
- [Background] Bonnet F, Marret E. Postoperative pain management and outcome after surgery. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):99-107. doi: 10.1016/j.bpa.2006.12.007. PMID 17489222
- [Background] Wong M, Morris S, Wang K, Simpson K. Managing Postoperative Pain After Minimally Invasive Gynecologic Surgery in the Era of the Opioid Epidemic. J Minim Invasive Gynecol. 2018 Nov-Dec;25(7):1165-1178. doi: 10.1016/j.jmig.2017.09.016. Epub 2017 Sep 28. PMID 28964926
- [Background] Griffith KC, Clark NV, Zuckerman AL, Ferzandi TR, Wright KN. Opioid Prescription and Patient Use After Gynecologic Procedures: A Survey of Patients and Providers. J Minim Invasive Gynecol. 2018 May-Jun;25(4):684-688. doi: 10.1016/j.jmig.2017.11.005. Epub 2017 Nov 14. PMID 29154933
- [Background] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Fuchs-Buder T, Meistelman C. [Monitoring of neuromuscular block and prevention of residual paralysis]. Ann Fr Anesth Reanim. 2009 Sep;28 Suppl 2:S46-50. doi: 10.1016/S0750-7658(09)72487-6. French. PMID 19887277
- [Background] Samimi S, Taheri A, Davari Tanha F. Comparison Between Intraperitoneal and Intravenous Lidocaine for Postoperative Analgesia After Elective Abdominal Hysterectomy, a Double-Blind Placebo Controlled Study. J Family Reprod Health. 2015 Nov;9(4):193-8. PMID 27047566
- [Background] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860
- [Background] Le Gall L, David A, Carles P, Leuillet S, Chastel B, Fleureau C, Dewitte A, Ouattara A. Benefits of intraoperative analgesia guided by the Analgesia Nociception Index (ANI) in bariatric surgery: An unmatched case-control study. Anaesth Crit Care Pain Med. 2019 Feb;38(1):35-39. doi: 10.1016/j.accpm.2017.09.004. Epub 2017 Oct 12. PMID 29033356
- [Background] Martini CH, Boon M, Bevers RF, Aarts LP, Dahan A. Evaluation of surgical conditions during laparoscopic surgery in patients with moderate vs deep neuromuscular block. Br J Anaesth. 2014 Mar;112(3):498-505. doi: 10.1093/bja/aet377. Epub 2013 Nov 15. PMID 24240315
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Background] Auquier P, Pernoud N, Bruder N, Simeoni MC, Auffray JP, Colavolpe C, Francois G, Gouin F, Manelli JC, Martin C, Sapin C, Blache JL. Development and validation of a perioperative satisfaction questionnaire. Anesthesiology. 2005 Jun;102(6):1116-23. doi: 10.1097/00000542-200506000-00010. PMID 15915023